CLINICAL TRIAL: NCT02567136
Title: A Longitudinal Study of Imaging Biomarkers in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Imaging Biomarkers in ALS
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 130126
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Amyotrophic Lateral Sclerosis: Patients with ALS
- Healthy Controls: Healthy control volunteers

SUMMARY:
The purpose of the study is to determine if we are able to find one or more biomarkers of Amyotrophic Lateral Sclerosis (ALS) and Primary Lateral Sclerosis (PLS) using magnetic resonance imaging (MRI) scans at different levels, 3 tesla (3T) and 7 tesla (7T). A biomarker is a measurable characteristic that can be used as an indicator of a particular disease state. Identifying biomarkers of a disease can lead to a better understanding of the disease as well as improved treatments. This study will enroll patients with ALS, PLS, and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 75 years of age inclusive.
* Willing and able to give signed informed consent that has been approved by the Institutional Review Board (IRB).

ALS patients:

* A clinical diagnosis of possible, laboratory-supported probable, probable, or definite ALS, according to a modified El Escorial criteria.

Exclusion Criteria:

* Diagnosis of other neurodegenerative diseases (Parkinson disease, Alzheimer disease, etc).
* Clinically significant history of unstable medical illness (unstable angina, advanced cancer, etc) over the last 30 days.
* Inability to undergo MRI scanning, including but not limited to unable to remain still in an MRI scanner for more than 30 minutes, claustrophobia, presence of paramagnetic substances or pacemakers in body, weight over 300 lbs, or in the opinion of the investigator, if there is a strong likelihood that the subject would not be able to lie flat comfortably for 75-90 minutes.
* The subject requires assistance to ambulate OR climb stairs, unless in the opinion of the investigator, and based upon the subject's rate of disease progression, the subject is likely to be able to participate in the MRI screening 12 months after enrollment.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll ALS patients seeking care at the University of Minnesota and age-matched healthy control volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2030-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Imaging biomarkers | 12 months
  Comparison of neurochemical concentrations and Diffusion Tensor Imaging (DTI) parameters between ALS subjects and age-matched normal subjects.

CONTACTS AND LOCATIONS:
Overall Officials: David Walk, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States